CLINICAL TRIAL: NCT01742546
Title: Effectiveness of Ultrasound Combine Transcutaneous Electrical Nerve Stimulation (TENS) in Treatment of Upper Trapezius Myofascial Pain: a Randomized Controlled Trial
Brief Title: Effectiveness of Ultrasound Combine TENS in Treatment of Upper Trapezius Myofascial Pain
Acronym: MPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sirindhorn National Medical Rehabilitation Centre (Other Government)
Responsible Party: Principal Investigator, Bootsakorn Loharjun, MD, Dr.Bootsakorn Loharjun, MD, Sirindhorn National Medical Rehabilitation Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SNMRC001
Record Dates: First submitted 2012-11-08; First posted 2012-12-05 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Myofascial Pain Syndromes
Keywords: myofascial pain syndrome; therapeutic ultrasound; combine therapy
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Therapeutic ultrasound combine TENS (Experimental): Use therapeutic ultrasound with simultaneous TENS for 10 minutes/session for 10 sessions/course.
  The therapeutic ultrasound machine in this study was Sonopuls 492 TM (Enraf-Nonius), this device has treatment head described by the manufacturers as having surface area as 5.8 cm2, ERA (Effective Radiating Area) of 5.0 cm2 and BNR (Beam Non-uniform Ratio) as max. 5.0. For electrotherapy unit which composes of 2 channels, output characteristics are constant current (CC) or constant voltage (CV), resolution of output signal is in steps of 0.2 mA and timer is limited to 30 minutes during ultrasound and combination therapy are operated.
  Interventions: Device: Therapeutic ultrasound combine TENS
- Therapeutic ultrasound with sham TENS (Sham Comparator): Use the same therapeutic ultrasound machine and place the electrode as experimental group but turn-off electrical current during treatment period
  Interventions: Device: Therapeutic ultrasound combine TENS

INTERVENTIONS:
Device: Therapeutic ultrasound combine TENS — Use ultrasound treatment parameters as continuous mode, 1 MHz in frequency and 1 w/cm2 for intensity and circular stroking of sound head over affected upper trapezius muscle throughout treatment period. For simultaneous TENS parameters as pulse frequency 100-150 pps, pulse duration 50- 80 µs and adjust amplitude as produce tingling for 10 minutes. The skin electrode should be placed near the active trigger in area of trapezius muscle. And the control group received sham TENS by turn-off electrical current.
  The therapeutic ultrasound machine in this study was Sonopuls 492 TM (Enraf-Nonius).
  Other Names: Therapeutic ultrasound combine simultaneous electrotherapy

SUMMARY:
To assess the effectiveness of therapeutic ultrasound combine transcutaneous electrical nerve stimulation (TENS) and therapeutic ultrasound in treatment of myofascial pain syndrome in upper trapezius muscle measured by mean change between pre and post treatment of pressure pain threshold (PPT), patient's complaint in pain intensity and the number of total tablet usage of acetaminophen in both groups.

DETAILED DESCRIPTION:
Myofascial pain syndrome (MPS) is one of the most common causes of musculoskeletal pain and can affect any skeletal muscles in the body.Myofascial pain is not fatal condition but it can significant reduced quality of life and is a major cause of time lost from work. There are various treatments, which divided into invasive and non-invasive therapies. In the recent clinical practice, there is a new type of combine treatment unit which composes of electrotherapy and ultrasound therapy in one unit. However, there is no conclusive evidence for supports the effectiveness of this combine therapy compare with the conventional ultrasound in treatment of myofascial pain especially in aspect of pain relief.

ELIGIBILITY:
Inclusion Criteria:

* Age > 20 years old
* Clinical diagnosis of myofascial trigger point pain at upper trapezius muscle(s) persisted more than 1 week but less than 6 months before recruitment time, first or recurrence episodes
* Baseline VAS more than or equal 4 at upper trapezius muscle

Exclusion Criteria:

* During the past 2 weeks had received injection or physical therapy at upper trapezius muscle or shoulder area
* Had experience of ultrasound combine transcutaneous electrical nerve stimulation (TENS)
* Had history of accidence or severe trauma to shoulder region
* Had serious musculoskeletal condition that need surgical intervention such as acute shoulder subluxation, abnormal neurological examination
* Insensate skin or sensory impairment around shoulder area
* Skin infection at shoulder area
* Had contraindication for U/S such as cardiac pacemaker, implantation, malignancy in relevant area, bleeding disorder, acute inflammatory musculoskeletal disease, pregnancy, lactation
* Unable to communication
* Unable to complete treatment session and follow protocol

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-06; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Evidence of pain relief by measured mean change between pre and post treatment of pressure pain threshold (PPT) | within two weeks or 10 times treatment-course
  pressure pain threshold (PPT) was measured with calibrated mechanical pressure algometer

SECONDARY OUTCOMES:
Evidence of pain relief by visual analogue scale(VAS) | within two weeks or 10 times treatment- course
  the patient's complaint in pain intensity which represent by mean change between pre and post treatment of visual analog scale

OTHER OUTCOMES:
Evidence of analgesic drug usage | within two weeks or 10 times treatment-course

CONTACTS AND LOCATIONS:
Overall Officials: Bootsakorn Loharjun, Medical Doctor, Principal Investigator — Sirindhorn National Medical Rehabilitation Centre
Locations (1):
- Sirindhorn National Medical Rehabilitation Centre, Muang, Changwat Nonthaburi, Thailand